CLINICAL TRIAL: NCT02928484
Title: Evaluación Del Efecto Del Suplemento Nutricional probiótico "Biopolis" Sobre la función Gastrointestinal
Brief Title: Evaluation of the Effect of a Probiotic Supplement Upon Gastrointestinal Function
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biopolis S.L. (Industry)
Collaborators: Hospital Universitario Central de Asturias (Other); National Research Council, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIEN-HUCA-IPLA
Record Dates: First submitted 2016-09-07; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Signs and Symptoms, Digestive; Dyspepsia
Keywords: Functional dyspepsia; Abdominal pain; Flatulence; Probiotics; Bifidobacterium; Lactobacillus
MeSH Terms: conditions — Signs and Symptoms, Digestive; Dyspepsia; Abdominal Pain; Flatulence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test product (Active Comparator): The volunteers, that have been randomly assigned to the Test product arm of the study, will be administered one oral capsule/day of the Probiotic mix CBP-004019/C (Biopolis SL) during the intervention period (1 month). The product contains 1X10Exp9 cfu/capsule of the probiotic mix (Bifidobacterium lactis, Bifidobacterium longum, Lactobacilus casei and Lactobacillus rhamnosus) plus maltodextrin and sugar.
  Interventions: Dietary Supplement: Probiotic mix CBP-004019/C
- Placebo product (Placebo Comparator): The volunteers that have been randomly assigned to this arm of the study will receive one oral capsule per day of the placebo product (Biopolis SL) during the 1 month intervention period. The product contains maltodextrin and sugar.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic mix CBP-004019/C — One capsule per day of the probiotic mix CBP-004019/C during one month.
  Arms: Test product
Dietary Supplement: Placebo — One capsule per day of the placebo (maltodextrin) during one month.
  Arms: Placebo product

SUMMARY:
The purpose of this pilot study is to evaluate whether a probiotic supplement improves gastrointestinal (GI) function.

DETAILED DESCRIPTION:
Sixty volunteers with functional GI disorders (Functional dyspepsia according to Rome-III criteria) will be recruited for a randomised, double-blind, placebo-controlled, two-arm parallel study in which the effect upon the gastrointestinal function of a probiotic mix containing bifidobacteria and lactobacilli (manufactured by Biopolis SL) will be compared with placebo (maltodextrin). The study design includes a 4 week run-in period, in which the volunteers will not consume any probiotics/prebiotics, followed by a 4 weeks intervention period (a daily capsule of placebo or probiotic) and an 8 weeks washout period. At the beginning/end of each period questionnaires in gastrointestinal function, dyspepsia related symptoms and diet will be carried out. A serum sample will be taken for cytokine levels determination. A faecal sample will be taken for 16S microbial population profiling and for determining the faecal levels of Bifidobacterium, Bacteriodes, Faecalibacterium, Akkermansia, Lactobacillus and Blautia by qPCR and the concentration of the main bacterial metabolites; acetate, propionate and butyrate by gas-chromatography.

ELIGIBILITY:
Inclusion Criteria:

* Functional dyspepsia (type postprandial distress or postprandial distress plus epigastric pain) diagnosed according to Rome III criteria

Exclusion Criteria:

* Celiac disease or other organic GI disease
* Orthorexia nervosa or other eating disorders
* Special dietary patterns (vegans, vegetarians, macrobiotic, exclusion diets, etc.)
* Extreme BMI (<18,8 or > 39,9)
* Metabolic disorders
* Positive Helicobacter pylori test
* Congenital IgA deficiency
* Lactose malabsorption/intolerance
* SIBO
* Diabetes
* Scleroderma, CREST, lupus or other connective tissue diseases
* Previous GI surgery or neoplastic disease
* Treatment with non steroidal anti-inflammatory drugs and/or acetyl salicylic acid.
* Pregnancy
* Menopause

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Functional dyspepsia symptoms | 3 months
  Physician determined symptoms according to Rome III criteria.

SECONDARY OUTCOMES:
Relative proportions of the main microbial groups of the intestinal microbiota | 3 months
  Global profile of intestinal microbiota composition established by 16S rRNA profiling
Dyspepsia associated quality of life | 3 months
  Questionaires for symptoms and QoL associated to dyspepsia and for anxiety/depression
Serum IFN-gamma levels | 3 months
  Determination of the serum concentration (pg/mL) of IFN-gamma
Serum TNF-alpha levels | 3 months
  Determination of the serum concentration (pg/mL) of TNF-alpha
Serum IL-12 levels | 3 months
  Determination of the serum concentration (pg/mL) of IL-12
Serum IL-4 levels | 3 months
  Determination of the serum concentration (pg/mL) of IL-4
Serum IL-10 levels | 3 months
  Determination of the serum concentration (pg/mL) of IL-10
Serum TGF-beta levels | 3 months
  Determination of the serum concentration (pg/mL) of TGF-beta
Fecal levels of Bifidobacterium | 3 months
  Determination of the levels (log cells/gr) of Bifidobacterium in fecal samples by qPCR
Fecal levels of Lactobacillus | 3 months
  Determination of the levels (log cells/gr) of Lactobacillus in fecal samples by qPCR
Fecal levels of Bacteroides | 3 months
  Determination of the levels (log cells/gr) of Bacteroides in fecal samples by qPCR
Fecal levels of Blautia | 3 months
  Determination of the levels (log cells/gr) of Blautia in fecal samples by qPCR
Fecal levels of Akkermansia | 3 months
  Determination of the levels (log cells/gr) of Akkermansia in fecal samples by qPCR
Fecal levels of Faecalibacterium | 3 months
  Determination of the levels (log cells/gr) of Faecalibacterium in fecal samples by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Suárez, MD, PhD, Principal Investigator — Hospital Universitario Central de Asturias, Servicio de Gastroenterología; Miguel Gueimonde, PhD, Principal Investigator — Consejo Superior de Investigaciones Científicas, IPLA-CSIC
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided